CLINICAL TRIAL: NCT07132177
Title: Targeted Naltrexone to Support Individuals Participating in Dry January
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000000
Record Dates: First submitted 2025-07-30; First posted 2025-08-20 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Misuse
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Naltrexone (Experimental): All participants will receive 31 pills of 50mg Naltrexone to take as needed over the month of January 2026
  Interventions: Drug: Naltrexone (oral tablets)

INTERVENTIONS:
Drug: Naltrexone (oral tablets) — All participants will receive 31 pills of 50 mg Naltrexone to take as needed over the month of January 2026.

SUMMARY:
This pilot open-label study will assess the feasibility, acceptability, and preliminary efficacy of targeted (as-needed) oral naltrexone in individuals participating in "Dry January," a month-long voluntary abstinence or reduction in alcohol use. Participants who do not meet criteria for alcohol use disorder (AUD) but are interested in reducing or abstaining from alcohol will receive a 31-day supply of 50mg oral naltrexone to take either prior to anticipated drinking or daily as a precaution. The study will evaluate recruitment, retention, adherence, and safety, as well as changes in alcohol use patterns, craving, mood, liver function, and quality of life. A qualitative interview at follow-up will explore participants' experiences using naltrexone during Dry January. Results will inform future randomized trials testing low-intensity, scalable interventions for non-treatment-seeking individuals seeking to reduce alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults aged 18 and above
* Intending to participate in "Dry January" in January of 2026 by either completely stopping or moderating (reducing) their drinking
* Available to travel to BWH CCI outpatient facilities for study visits

Exclusion Criteria:

* DSM-5 diagnosis of moderate or severe AUD
* Seeking treatment for AUD
* Currently receiving medications for treating AUD (naltrexone, acamprosate, disulfiram)
* CIWA score > 3 at the time of enrollment
* Blood alcohol level (BAL) > 0 at enrollment
* Current DSM-5 diagnosis of any other SUD except for tobacco use disorder
* History of any inpatient alcohol withdrawal (i.e. "detox") admission
* History of severe withdrawal syndrome including withdrawal seizure or delirium tremens
* Active psychosis, mania, suicidality or homicidally or any psychiatric condition that impair ability to provide informed consent
* Liver function test greater than 3 times upper normal limit or severe renal impairment
* History of hypersensitivity or allergy to naltrexone
* Currently or anticipating requiring opioid analgesics for pain during the trial
* Pregnant or breastfeeding
* Anticipated to permanently leave the Boston area during the duration of the trial.
* Anticipated to be enrolled in another clinical drug trial during participation of this trial
* Any other reason or clinical condition that the investigators judge may interfere with study participation and/or be unsafe for a participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | Up to 3 business days following baseline visit
  Recruitment: Proportion of those screened who successfully enroll in the trial. Greater than 75% enrollment will be considered excellent, and greater than 50% enrollment will be considered good.
Retention feasibility | Up to 3 business days following baseline visit
  Proportion of those enrolling who successfully complete all study visits. Greater than 80% retention will be considered excellent, and greater than 70% retention will be considered good.
Intervention acceptability | Up to 3 business days following baseline visit
  The 4-item Acceptability of Intervention Measure (AIM) will be used, measured on a 5-point scale.
Naltrexone adherence | 1 month during the month of Januaray 2026
  The total number of naltrexone tablets taken will be assessed by pill count.
Safety Measure | Up to 3 business days following baseline visit
  The incidence and severity of adverse events (AEs) will be documented using the Patient Rated Inventory of Side Effects (PRISE)6: A self-report tool to qualify side effects. For each domain, the patient rates whether the symptoms are tolerable or distressing.

SECONDARY OUTCOMES:
Change in Overall Drinking | Up to 3 business days following baseline visit
  Drinks per drinking days (DDD) will be calculated using the Time-Line Follow Back (TLFB)7, a gold-standard method of evaluating substance use. The TLFB results will also calculate proportion of heavy drinking days and proportion of days abstinent during the 4-week intervention.
Alcohol Withdrawal | Up to 3 business days following baseline visitn
  Clinical Institute Withdrawal Assessment (CIWA)8: Tool for assessing alcohol withdrawal.
Quality of Life Assessment | Up to 3 business days following baseline visit
  WHO Quality of Life (WHOQOL-BREF)71: A 26-item quality of life scale.
Alcohol Craving | Up to 3 business days following baseline visit
  Penn Alcohol Craving Scale:13 A measure of craving for alcohol.
Overall Alcohol Consumption | Up to 3 business days following baseline visit
  PEth: An alcohol biomarker to assess overall alcohol consumption of the prior 2-4 weeks.
Medication Adherence | 1 month during the month of January 2026
  Morisky Medication Adherence Scale-MMAS: a 4 item self-report tool designed to assess how well patients stick to their prescribed medication regimens.
Acceptability of Intervention | Up to 3 business days following baseline visit
  Acceptability of Intervention Measure (AIM): 4 item scale
Safety Check | Up to 3 business days following baseline visit
  Liver Function Test: lab work/blood test

OTHER OUTCOMES:
Interview Outcomes | At final study visit
  A qualitative interview at follow-up will explore participants' experiences using naltrexone during Dry January.

CONTACTS AND LOCATIONS:
Overall Officials: Joji Suzuki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No